CLINICAL TRIAL: NCT04187313
Title: Increasing Notifications of Tuberculosis From Private Practitioners: A Randomised Controlled Trial
Brief Title: Increasing Notifications of Tuberculosis From Private Practitioners
Acronym: INSTEP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Collaborators: University of Otago (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Panji Fortuna Hadisoemarto, MD, MPH, Universitas Padjadjaran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TB-201911.02
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Public-Private Sector Partnership; Mobile Applications
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: The intervention will be administered to private practitioners in the selected areas (clusters), at their place of practice. Once the study participants have received the intervention, real-time monitoring of referral practice of patients for diagnosis and notification will be undertaken through the web-link to the app.
Who Masked: Outcomes Assessor
Masking Description: Study statistician will not be aware of intervention assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm will comprise study participants who receive intervention package (i.e. private practitioners in the selected areas who agree to participate).
  Interventions: Other: INSTEP2 intervention package
- Control (No Intervention): Private practitioners in the control areas will receive no intervention.

INTERVENTIONS:
Other: INSTEP2 intervention package — The Intervention will comprise: An electronic notification system, a standardized education about the signs and symptoms of TB and TB management and an individualised plan for each PP with respect to their approach to the diagnosis and management of TB suspects.
  The electronic system is a refinement of the electronic referral and report-back system using a mobile phone 'app'. The system will enable essential data to be uploaded, consistent with National TB Control Programme forms.
  The education package will be focused on TB suspect identification, provisional diagnosis and referral, including how to use the mobile phone 'app'. We will also develop a simple individualised approach for the management of TB suspects, which takes into account the context around each PP's practice, identifying the most efficient and feasible approach to obtaining a diagnosis and notifying TB patients.
  Arms: Intervention

SUMMARY:
Tuberculosis (TB) is the third leading cause of death in Indonesia. Disturbingly, the prevalence survey showed that over half of TB cases in Indonesia are not notified. The huge private sector in Indonesia, comprising an estimated 70,000 practitioners, provides over 50% of health care but notifies less than 10% of all diagnosed TB cases.

INSTEP2 is a cluster randomised controlled intervention trial. The multi-component public health intervention will be administered to private practitioners (PP) in Community Health Centre (CHC) clusters. The change in the number of TB notifications over 12 months before, and 12 months after, the intervention will be compared between study arms. Hypothesis related to the Primary Efficacy Endpoint: A tailored intervention in PPs will increase TB notifications.

DETAILED DESCRIPTION:
As part of advancing Public-Private Mix (PPM), the government made TB notification mandatory in 2016, but intervention is likely to be needed for notifications to increase substantially. Such intervention needs to be based on a sound understanding of contextual factors around PPs and how they relate to the public sector with respect to the diagnosis, treatment and reporting of TB cases.

This is a cluster randomised controlled trial of a multi-component public health intervention to increase notifications of TB from PPs in Bandung, Indonesia. Clusters are CHC areas and the intervention will be administered directly to PPs in sub-districts randomised to the intervention arm. The CHCs in both arms will be informed about the study and asked, through the National TB Control Programme, to make their notification data available and their willingness will be recorded. No intervention will be given to PPs in the control arm. Notifications will be obtained directly from routine records, with accompanying information gathered about the address of the patient and referring doctor. Notified TB cases are, by definition, TB cases who have been commenced on TB treatment, noting that some referred 'TB cases' will be diagnosed as not having TB by CHC staff.

The intervention will be administered to PPs in areas around 15 CHCs (clusters), at their place of practice. PPs in the control areas will receive no intervention. The intervention will comprise: (1) An electronic referral and notification system; (2) Education about signs and symptoms of TB and TB management; (3) An individualised practitioner plan for diagnostic and management pathways.

The primary endpoint is the change in the number of notifications of TB from the 12 months before to the 12 months after the intervention is fully implemented. This change in the number of notifications will be compared between intervention clusters and control clusters.

Safety oversight by a Data and Safety Monitoring Board (DSMB) will not be required for this public health intervention trial. However, an internal Data Monitoring Committee (DMC) will be established to oversee the study, focused on data quality. A quality management plan will be developed to describe a site's quality management. Quality control (QC) procedures will be implemented beginning with the data entry system and data QC checks that will be run on the database will be automatically generated on a weekly basis and any quality issues identified will be reviewed by the DMC and a plan put in place for resolution. Following written Standard Operating Procedures (SOPs), visiting investigators will verify that the trial is conducted and data are generated, documented (recorded), and reported in compliance with the protocol. The investigational site will provide direct access to all source data/documents, and reports for the purpose of the verification visits.

ELIGIBILITY:
Inclusion Criteria:

* All medically qualified private practitioners (PPs) in the intervention arm who reported having diagnosed at least one TB case in the past 3 months
* Intend to work in the current location for the duration of the study as their primary place of private practice

Exclusion Criteria:

* Unable to use an electronic device for referral/notification
* More than 3 months of non-practice during the study period is anticipated
* They are not a qualified medical practitioner, with the appropriate medical authority in Indonesia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Increased notification of tuberculosis (TB) by study participants | 12 months before to the 12 months after the intervention
  Increased notifications of TB by private practitioners in Bandung, Indonesia

SECONDARY OUTCOMES:
Proportion of referred patients in the intervention and control arms that are actually diagnosed with TB | 12 months before to the 12 months after the intervention
  Proportion of referrals from private practitioners that are actually diagnosed with TB (i.e. bacteriologically confirmed TB)
Restricted analysis of primary outcome | 12 months before to the 12 months after the intervention
  Analysis of the primary outcome, limited to notifications of patients who live in the Community Health Center (CHC) area where they are notified

CONTACTS AND LOCATIONS:
Overall Officials: Philip Hill, Professor, Principal Investigator — University of Otago
Locations (1):
- Universitas Padjadjaran Teaching Hospital, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahendradhata Y, Lestari T, Probandari A, Indriarini LE, Burhan E, Mustikawati D, Utarini A. How do private general practitioners manage tuberculosis cases? A survey in eight cities in Indonesia. BMC Res Notes. 2015 Oct 14;8:564. doi: 10.1186/s13104-015-1560-7. PMID 26468010
- [Background] Irawati SR, Basri C, Arias MS, Prihatini S, Rintiswati N, Voskens J, Kimerling ME. Hospital DOTS linkage in Indonesia: a model for DOTS expansion into government and private hospitals. Int J Tuberc Lung Dis. 2007 Jan;11(1):33-9. PMID 17217127
- [Background] Surya A, Setyaningsih B, Suryani Nasution H, Gita Parwati C, Yuzwar YE, Osberg M, Hanson CL, Hymoff A, Mingkwan P, Makayova J, Gebhard A, Waworuntu W. Quality Tuberculosis Care in Indonesia: Using Patient Pathway Analysis to Optimize Public-Private Collaboration. J Infect Dis. 2017 Nov 6;216(suppl_7):S724-S732. doi: 10.1093/infdis/jix379. PMID 29117347
- [Background] Probandari A, Utarini A, Hurtig AK. Achieving quality in the Directly Observed Treatment Short-course (DOTS) strategy implementation process: a challenge for hospital Public-Private Mix in Indonesia. Glob Health Action. 2008 Dec 17;1. doi: 10.3402/gha.v1i0.1831. PMID 20027243
- [Background] Reviono R, Setianingsih W, Damayanti KE, Ekasari R. The dynamic of tuberculosis case finding in the era of the public-private mix strategy for tuberculosis control in Central Java, Indonesia. Glob Health Action. 2017;10(1):1353777. doi: 10.1080/16549716.2017.1353777. PMID 28766465
- [Background] Lestari BW, Arisanti N, Siregar AYM, Sihaloho ED, Budiman G, Hill PC, Alisjahbana B, McAllister S. Feasibility study of strengthening the public-private partnership for tuberculosis case detection in Bandung City, Indonesia. BMC Res Notes. 2017 Aug 14;10(1):404. doi: 10.1186/s13104-017-2701-y. PMID 28807020
- [Background] Lei X, Liu Q, Escobar E, Philogene J, Zhu H, Wang Y, Tang S. Public-private mix for tuberculosis care and control: a systematic review. Int J Infect Dis. 2015 May;34:20-32. doi: 10.1016/j.ijid.2015.02.015. Epub 2015 Feb 23. PMID 25722284
- [Background] Artawan Eka Putra IW, Utami NW, Suarjana IK, Duana IM, Astiti CI, Putra IW, Probandari A, Tiemersma EW, Wahyuni CU. Factors associated to referral of tuberculosis suspects by private practitioners to community health centres in Bali Province, Indonesia. BMC Health Serv Res. 2013 Oct 28;13:445. doi: 10.1186/1472-6963-13-445. PMID 24165352
- See also: World Health Organisation. PPM DOTS in Indonesia: a strategy for action — https://apps.who.int/iris/handle/10665/68349

DOCUMENTS (2):
  • Study Protocol (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/13/NCT04187313/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT04187313/SAP_001.pdf